CLINICAL TRIAL: NCT03274115
Title: BLI (Blue Light Imaging) Application for the Histological Characterization of Colorectal Polyps
Brief Title: BLI (Blue Light Imaging) for the Histological Characterization of Colorectal Polyps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valduce Hospital (Other)
Responsible Party: Principal Investigator, Franco Radaelli, MD, Head of Gastrointestinal Endoscopy Unit, Valduce Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 341/2017 bis
Record Dates: First submitted 2017-08-29; First posted 2017-09-06 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Adenoma Colon

STUDY DESIGN:
Intervention Model Description: Patients with at least one polyp <1 cm in size will be randomized in two groups. In the Group 1 (White Light Group), all polyps <10mm will be evaluated with white light and prediction of histology (hyperplastic versus adenomatous) will be made. In the Group 2 (BLI Group) , all polyps <10mm in size will be evaluated with BLI and scored as hyperplastic (type 1) or adenomatous (type 2) by applying the NICE ( Narrow-band Imaging International Colorectal Endoscopic) classification. The level of endoscopist's confidence in predicting real-time histology (high or low confidence) for any polyp will be also recorded.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- White Light (WL) (No Intervention): White light will be used for histology prediction of colonic polyps (hyperplastic versus adenomatous).
- Blue Light Imaging (BLI) (Active Comparator): Switch from white light to BLI (Blue Laser Imaging) to predict the histology of colonic polyps.
  Interventions: Device: BLI (Blue Laser Imaging)

INTERVENTIONS:
Device: BLI (Blue Laser Imaging) — Switch from white light to BLI (Blue Laser Imaging) to predict the histology of colonic polyps
  Arms: Blue Light Imaging (BLI)

SUMMARY:
The accuracy of real-time histology prediction (hyperplastic vs. adenomas) of colonic polyps using white light high-definition endoscopes is suboptimal. Blue laser imaging (BLI) is a new system for image-enhanced endoscopy using laser light, that is incorporated in the last generation Fuji high- definition videocolonscopes ELUXEO. Blue laser imaging (BLI) utilizes two monochromatic lasers instead of xenon light: a 410 nm laser visualizes vascular microarchitecture, similar to narrow band imaging, and a 450 nm laser provides white light by excitation.This system should enhance the microvascular pattern of superficial lesions, making the histological prediction easier.

Aim of the study is to compare the accuracy of white light and BLI systems in real-time histology prediction of colonic polyps.

For this purpose all colonscopies will be performed in a standard fashion using white light. When a polyps <10mm in size will be identified, patients will be randomized in two groups. In the Group 1 (White Light Grroup), all polyps <10mm will be evaluated with white light and prediction of histology (hyperplastic versus adenomatous) will be made by means of white light. In the Group 2 (BLI Group) , all polyps <10mm in size will be evaluated with BLI and scored as hyperplastic (type 1) or adenomatous (type 2) by applying the NICE (Narrow-band Imaging International Colorectal Endoscopic) classification, indicating color/vessel/surface pattern. The level of endoscopist's confidence in predicting histology (high or low confidence) for any polyp will be also recorded.

Diagnostic performances of the endoscopists (sensitivity, specificity, positive and negative predictive values) will be calculated comparing endoscopist's prediction and pathology report, considered as reference standard in both study groups in order to evaluate the accuracy of real-time histology prediction by using BLI or white light.

ELIGIBILITY:
Inclusion Criteria:

* All outpatients referred for colonoscopy

Exclusion Criteria:

* inadequatete bowel preparation (Boston Bowel Preparation Scale (BBPS) < 2 in one colonic segment)
* previous colonic resection
* inflammatory bowel disease
* ereditary polyposic syndromes
* patients on antithrombotics precluding polyp resection
* absence of informed consent
* inpatients or patients undergoing urgent colonscopy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic performances (sensitivity, specificity, positive and negative predictive values) in predicting colonic polyp histology | one year
  Diagnostic performances (sensitivity, specificity, positive and negative predictive values) in predicting colonic polyp histology will be calculated comparing endoscopist's prediction with pathology result (reference standard).

CONTACTS AND LOCATIONS:
Overall Officials: Franco Radaelli, Principal Investigator — Valduce Hospital
Locations (1):
- Gastroenterology Unit, Valduce Hospital, Como, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rondonotti E, Paggi S, Amato A, Mogavero G, Andrealli A, Conforti FS, Conte D, Spinzi G, Radaelli F. Blue-light imaging compared with high-definition white light for real-time histology prediction of colorectal polyps less than 1 centimeter: a prospective randomized study. Gastrointest Endosc. 2019 Mar;89(3):554-564.e1. doi: 10.1016/j.gie.2018.09.027. Epub 2018 Sep 28. PMID 30273590